CLINICAL TRIAL: NCT01071811
Title: The Effect After 12 Weeks of Having Received a Pedometer and a Pedometer Program on Physical Activity, Health Measurements, Self-rated Health, Stress, and Sleep Quality: a Randomized Controlled Trial
Brief Title: The Effect After 12 Weeks of Having Received a Pedometer and a Pedometer Program on Physical Activity and Health
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Morten Grønbæk, National Institut of Public Health, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1975
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Physical Inactivity
Keywords: Randomized controlled trial; Pedometer; Physical activity; Health measurement; Self-rated health; Stress; Sleep quality
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Sleep Initiation and Maintenance Disorders | interventions — Randomized Controlled Trials as Topic; Health; Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Participants assigned to the control group received a leaflet from the National Board of Health in Denmark recommending all adults to be physical active for 30 minutes each day of moderate intensity.
  Interventions: Behavioral: Pedometer-based intervention
- Pedometer group (Experimental): Received a pedometer (Yamax Digi-Walker SW-200), a book with a pedometer program, a handout with a summary of the pedometer program, and a calendar for registration of daily steps.
  Interventions: Behavioral: Pedometer-based intervention

INTERVENTIONS:
Behavioral: Pedometer-based intervention — The participants were randomly assigned to either a pedometer group or a control group by drawing a sealed envelope with a unique randomizing number. The participants in the pedometer group received a pedometer (Yamax Digi-Walker SW-200), a book with a pedometer program(18), a handout with a summary of the pedometer program, and a calendar for registration of daily steps. During the trial period they were asked to reset the pedometer every morning and to wear it during the entire day. In the evening they should take the pedometer off and register the accumulated steps in the calendar. After three, six, and nine weeks, the participants in the pedometer group got a mail to encourage them to keep using the pedometer and follow the program.
  Other Names: Randomized controlled trial; Pedometer; Pedometer program; Health; Self-rated health; Stress; Sleep

SUMMARY:
Physical activity is associated with a reduced risk of several chronic diseases in addition to all-cause mortality. Hence for public health purposes, knowledge of effective interventions to increase the physical activity level in the population is important.

The objective of this randomized controlled trial was to examine the effect 12 weeks after having received a pedometer and a pedometer program on physical activity, health measurements, self-rated health, stress, and sleep quality.

A total of 223 men and 445 women were randomly assigned to either a pedometer group (n = 333) in which participants received a pedometer and pedometer program or a control group (n = 335). Of the participants included in the study 198 and 178 completed the health examination, and 192 and 187 completed the questionnaire at follow up in the pedometer group and in the control group, respectively.

DETAILED DESCRIPTION:
The results from the KRAM Study are used as baseline for this intervention. In the KRAM study all adult citizens (18+ years) in 13 Danish municipalities were invited by letter to take part in an internet based questionnaire concerning socio-demography, life style, and other health aspects. Furthermore, a random sample of the citizens was invited to participate in a health examination. A total of 76.484 of the invited 538.497 citizens filled in the entire or partially the questionnaire and 18.065 of the invited 180.103 citizens completed the health examination. The examination included the following measurements: Blood pressure, height, weight, fat percentage, blood samples, pulmonary function, bone mineral density, muscle strength, balance test, and aerobic fitness.

Intervention The intervention was carried out in three of the 13 municipalities (Silkeborg, Frederiksberg, and Varde). Participants with a low aerobic fitness (defined for men and women in different age groups) or those who reported being sedentary or light physically active in leisure time were - after they had accomplished the health examination - invited to participate in the intervention. Participants were not included if they participated in other interventions initiated in relation with the KRAM Study or if they were pregnant. All participants gave informed consent. The protocol was approved by the Scientific Ethical Committee B for the Capital Region of Denmark (H-B-2008-097).

The participants were randomly assigned to either a pedometer group or a control group by drawing a sealed envelope with a unique randomizing number. The participants in the pedometer group received a pedometer (Yamax Digi-Walker SW-200), a book with a pedometer program, a handout with a summary of the pedometer program, and a calendar for registration of daily steps. The aim of the program is to guide people to use a pedometer and increase their steps with 20 % each week until they reach their goal. During the trial period, they were asked to reset the pedometer every morning and to wear it during the entire day. In the evening, they should take the pedometer off and register the total number of steps in the calendar. After three, six, and nine weeks, the participants in the pedometer group got a mail to encourage them to keep using the pedometer and follow the program. Participants assigned to the control group received a leaflet from the National Board of Health in Denmark recommending all adults to be physical active for 30 minutes each day of moderate intensity.

Follow up After 12 weeks, participants were invited by letter to answer a short questionnaire. Furthermore, they were invited to participate in a health examination including the measurements of blood pressure, weight, fat percentage, and aerobic fitness. The researchers who performed the examinations were blinded to group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Low aerobic fitness (defined for men and women in different age groups)
* Reported being sedentary or light physically active in leisure time

Exclusion Criteria:

* Participated in other interventions initiated in relation with the KRAM Study
* Were pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Physical activity (walking time, sitting time, physical activity level in leisure time) | 12 weeks

SECONDARY OUTCOMES:
Health measurements (blood pressure, weight, fat percentage, and aerobic fitness), self-rated health, stress, and sleep quality | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Morten Grønbæk, professor, Study Director — National Institut of Public Health, University of Southern Denmark
Locations (3):
- Denmark (3):
  - The municipiality of Frederiksberg, Frederiksberg
  - The municipiality of Silkeborg, Silkeborg
  - The municipiality of Varde, Varde

REFERENCES:
- [Derived] Petersen CB, Severin M, Hansen AW, Curtis T, Gronbaek M, Tolstrup JS. A population-based randomized controlled trial of the effect of combining a pedometer with an intervention toolkit on physical activity among individuals with low levels of physical activity or fitness. Prev Med. 2012 Feb;54(2):125-30. doi: 10.1016/j.ypmed.2011.12.012. Epub 2011 Dec 19. PMID 22200586